CLINICAL TRIAL: NCT00226291
Title: The Clinical Informationist: Does the Model Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nunzia Giuse, Assistant Vice Chancellor for Knowledge Management; Director, Eskind Biomedical Library; Professor, Department of Biomedical Informatics, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 040624; 5R01LM007849 (NIH)
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Critical Illness
Keywords: EBM; evidence based medicine; informationist; clinical medical librarian
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synthesized evidence report (Experimental): Each consultation response included a documented bibliographic search strategy with corresponding references, a targeted list of full-text articles, and a written synthesis and critique of the relevant research materials.
  Interventions: Other: Synthesized evidence report
- No evidence report (No Intervention)

INTERVENTIONS:
Other: Synthesized evidence report — Each consultation response included a documented bibliographic search strategy with corresponding references, a targeted list of full-text articles, and a written synthesis and critique of the relevant research materials.
  Other Names: Literature summary; Evidence report
  Arms: Synthesized evidence report

SUMMARY:
This study is investigating the effects of an established clinical informationist program (evidence-based practice support service in which information professionals with significant clinical knowledge bases and advanced information seeking and appraisal skills) on clinical decision making at selected critical care units at Vanderbilt University Medical Center

DETAILED DESCRIPTION:
Background To evaluate the role of the Clinical Informatics Consult Service(CICS), an informationist service at the Eskind Biomedical Library (EBL) at Vanderbilt University Medical Center (VUMC, in clinical decision-making, the EBL has been awarded a 3-year grant from the National Library of Medicine (5 R01 LM07849-02). The CICS is a well-established program that facilitates evidence-based practice by delivering targeted information in answer to complex, patient-specific questions. The CICS places librarians with specialized training in medical subject areas and in information retrieval ("clinical informationists") on clinical teams in intensive care settings. Acting as expert consultants, they analyze the biomedical literature to identify, filter, and present the best examples of each clinical viewpoint expressed about key problems.

Evaluation Project Working in cooperation with the Center for Evaluation and Program Improvement (CEPI) at Peabody College of Vanderbilt, the investigators will evaluate formally the role of CICS in clinical decision-making and evidence-seeking behavior. While past studies have evaluated clinical medical librarians' roles, few if any studies have examined the effectiveness and utility of the new clinical informationist approach in sites where informationists are well-established.

The project will also create reusable evaluation tools transferable across environments. Through a combination of observation and interviews, investigators will examine librarian involvement in three existing Vanderbilt CICS intensive care units. The project will collect detailed information about the ways in which clinicians incorporate CICS-provided information into their workflows. Next, investigators will conduct a randomized trial to evaluate the effect of CICS on decision-making. Investigators will compare clinicians' intended course of care vs. actual care when CICS results are provided and when clinicians seek information themselves.

Finally, "virtual cases" developed from actual patient CICS-related scenarios in each clinical unit will be incorporated into training tools that can be used to export elements of the CICS model to other locations. Demonstration of the utility of the clinical informationist approach can foster widespread adoption nationally, and increase the degree to which clinical practice becomes evidence-based.

ELIGIBILITY:
Inclusion Criteria:

Evidence-based questions requested by clinician on current service as an attending, resident, fellow, or nurse practitioner on one of the units included in the study

Exclusion Criteria:

All others

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2004-08; Primary Completion 2006-02 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Immediate and potential future clinical decisions | 3 days post-consult

SECONDARY OUTCOMES:
Clinical action index | 3 days post-consult
Number of research articles read | 3 days post-consult
Satisfaction | 3 days post-consult
Colleague consults | 3 days post-consult
Time spent searching the literature | 3 days post-consult

CONTACTS AND LOCATIONS:
Overall Officials: Nunzia B Giuse, MD, MLS, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Giuse NB, Koonce TY, Jerome RN, Cahall M, Sathe NA, Williams A. Evolution of a mature clinical informationist model. J Am Med Inform Assoc. 2005 May-Jun;12(3):249-55. doi: 10.1197/jamia.M1726. Epub 2005 Jan 31. PMID 15684125
- [Background] Rosenbloom ST, Giuse NB, Jerome RN, Blackford JU. Providing evidence-based answers to complex clinical questions: evaluating the consistency of article selection. Acad Med. 2005 Jan;80(1):109-14. doi: 10.1097/00001888-200501000-00025. PMID 15618105
- [Background] Jerome RN, Giuse NB, Gish KW, Sathe NA, Dietrich MS. Information needs of clinical teams: analysis of questions received by the Clinical Informatics Consult Service. Bull Med Libr Assoc. 2001 Apr;89(2):177-84. PMID 11337949
- [Background] Florance V, Giuse NB, Ketchell DS. Information in context: integrating information specialists into practice settings. J Med Libr Assoc. 2002 Jan;90(1):49-58. PMID 11838460
- [Background] Giuse NB, Kafantaris SR, Miller MD, Wilder KS, Martin SL, Sathe NA, Campbell JD. Clinical medical librarianship: the Vanderbilt experience. Bull Med Libr Assoc. 1998 Jul;86(3):412-6. No abstract available. PMID 9681179
- [Background] Giuse NB. Advancing the practice of clinical medical librarianship. Bull Med Libr Assoc. 1997 Oct;85(4):437-8. No abstract available. PMID 9431437
- [Background] Sathe NA, Todd P, Gregg W, Clark J, Giuse NB. Virtual cases as a tool to promote the incorporation of EBM techniques into housestaff training . Medical Library Association Annual Meeting, Phoenix, AZ, May 2006. (Poster)
- [Result] Mulvaney SA, Bickman L, Giuse NB, Lambert EW, Sathe NA, Jerome RN. A randomized effectiveness trial of a clinical informatics consult service: impact on evidence-based decision-making and knowledge implementation. J Am Med Inform Assoc. 2008 Mar-Apr;15(2):203-11. doi: 10.1197/jamia.M2461. Epub 2007 Dec 20. PMID 18096918
- [Result] Mulvaney S, Bickman L, Lambert W, Sathe N, Jerome R, Guise NB. Barriers to and facilitators of evidence based practices in physicians. Society for Behavioral Medicine 28th Annual Meeting. Washington, DC. March 2007. (Poster)